CLINICAL TRIAL: NCT03049592
Title: High-risk Obstetrical Patient Intervention to Promote Birth Interval Spacing Utilizing the Contraceptive CHOICE Project Script to Reduce Unintended Subsequent Pregnancies
Brief Title: High-risk Obstetrical Patient Intervention Utilizing the Contraceptive CHOICE Project Script
Acronym: HIBISCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160020
Record Dates: First submitted 2016-11-23; First posted 2017-02-10 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Diabetes; Contraception
Keywords: Diabetes; Contraception; Prenatal Counseling
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIBISCUS counseling (Experimental): Subject receives a third trimester prenatal appointment with a family planning specialist for contraceptive counseling (utilizing the Contraceptive CHOICE counseling script emphasizing the WHO birth-to-pregnancy recommendation of 18 months) and a follow up postpartum contraception visit with a family planning specialist.
  Interventions: Other: HIBISCUS counseling
- Standard counseling (No Intervention): Subect receives standard high-risk prenatal care and postpartum contraception provision by the referring community clinic. The community clinic offer standard family planning counseling that does not emphasize utilizing of long-acting reversible contraception to promote birth-to-pregnancy spacing of 18 months. This scenario is current the standard practice at the institutions.

INTERVENTIONS:
Other: HIBISCUS counseling — Third trimester prenatal appointment with a family planning specialist for contraceptive counseling utilizing the Contraceptive CHOICE counseling script - emphasizing the WHO birth-to-pregnancy recommendation of 18 months, and a follow up postpartum contraception visit with a family planning specialist.
  Arms: HIBISCUS counseling

SUMMARY:
High-risk obstetrical patient Intervention to promote Birth Interval Spacing utilizing the Contraceptive CHOICE project script to reduce Unintended Subsequent pregnancies (HIBISCUS) is a collaborative study utilizing qualitative methods to assess the acceptability including a family planning specialist's postpartum contraception counseling during and after prenatal care among Latina obstetric women with pre-gestational diabetes. The investigators will compare the effectiveness of HIBISCUS versus usual contraceptive counseling on Long-Acting Reversible Contraception (LARC) use at 3 months postpartum.

DETAILED DESCRIPTION:
The purpose of this research is to address this gap in long-acting reversible contraception (LARC) counseling among Latinas who have pregnancies complicated by pre-gestational diabetes in order to promote optimal birth-to-pregnancy spacing and planned pregnancies with optimal glucose control. The investigators will utilize Contraceptive CHOICE project which was LARC focused counseling script and removed the cost of contraception. This study had a LARC utilization of 75% compared to the national use of LARC of 7.2% The investigators will conduct a pilot randomized controlled trial among Latina obstetrics patients with pre-gestational diabetes involving a prenatal and postpartum visit with a family planning specialist versus usual contraceptive counseling. The family planning specialist counseling will utilize the Contraceptive CHOICE Project script promoting LARC, 18 month birth-to-pregnancy recommendation and preconception counseling. The intervention's name is HIBISCUS.

ELIGIBILITY:
Inclusion Criteria:

* Latina obstetric women
* Pre-gestational diabetes
* Obtaining prenatal care in the high-risk obstetrical clinic - Diabetes in Pregnancy

Exclusion Criteria:

* Desires sterilization

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Utilization of LARC | 1 year
  Utilization of LARC postpartum

SECONDARY OUTCOMES:
Acceptability of contraceptive counseling intervention by patients and clinicians | 1 year
  Comparison of rates and reasons for acceptance vs. non-acceptance of contraceptive counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD MPH, Principal Investigator — UC San Diego Health System
Locations (1):
- UC San Diego Health System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peipert JF, Madden T, Allsworth JE, Secura GM. Preventing unintended pregnancies by providing no-cost contraception. Obstet Gynecol. 2012 Dec;120(6):1291-7. doi: 10.1097/aog.0b013e318273eb56. PMID 23168752
- [Background] Daniels K, Daugherty J, Jones J. Current contraceptive status among women aged 15-44: United States, 2011-2013. NCHS Data Brief. 2014 Dec;(173):1-8. PMID 25500343
- [Background] World Health Organization. Report of a WHO Technical Consultation on Birth Spacing, Geneva, Switzerland, June 13-15, 2005. Report Geneva, Switzerland: World Health Organization, 2006.
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Thiel de Bocanegra H, Chang R, Howell M, Darney P. Interpregnancy intervals: impact of postpartum contraceptive effectiveness and coverage. Am J Obstet Gynecol. 2014 Apr;210(4):311.e1-311.e8. doi: 10.1016/j.ajog.2013.12.020. Epub 2013 Dec 13. PMID 24334205
- [Background] Hardy E, Santos LC, Osis MJ, Carvalho G, Cecatti JG, Faundes A. Contraceptive use and pregnancy before and after introducing lactational amenorrhea (LAM) in a postpartum program. Adv Contracept. 1998 Mar;14(1):59-68. doi: 10.1023/a:1006527711625. PMID 9587009